CLINICAL TRIAL: NCT04644874
Title: Predictive Value of Geriatric Oncology Screening and Geriatric Assessment in Older Patients With Solid Cancers: A Prospective G8 Study
Brief Title: Geriatric Oncology Screening of Older Patients With Solid Cancers
Acronym: PROGNOSIS-G8
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Academy of Geriatric Cancer Research (Unknown); Danish Cancer Society (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Helena Ditzel, Principal Investigator, Odense University Hospital
Other Study IDs: PROGNOSIS-G8; R247-A14382 (Other Grant/Funding Number: Danish Cancer Society); 20/ 17768 (Other: Region of Southern Denmark)
Record Dates: First submitted 2020-11-12; First posted 2020-11-25 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Solid Carcinoma; Frailty; Age; Geriatrics; Screening; Cancer
Keywords: Older adults; Cancer patients; Neoplasms; Frailty; Comprehensive geriatric assessment; Geriatric screening; Geriatric 8; modified Geriatric 8; G8; mG8; elderly; screening
MeSH Terms: conditions — Frailty; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older cancer patients: All outpatients, age 70 years or more, with solid malignancies, referred to the Department of Oncology at Odense University Hospital for 1st line antineoplastic treatment or information,
  Interventions: Diagnostic Test: Geriatric 8; Diagnostic Test: modified Geriatric 8; Diagnostic Test: 30 second chair stand test; Diagnostic Test: Handgrip Strength Test

INTERVENTIONS:
Diagnostic Test: Geriatric 8 — The G8 is an eight-item screening tool, developed for older cancer patients. The G8 score ranges from 0 (heavily impaired) to 17 (not at all impaired), with a cut-off for potential frailty of ≤14.
  Other Names: G8
Diagnostic Test: modified Geriatric 8 — The mG8 is a modified version of the Geriatric 8 screening tool, consisting of 6-items. The mG8 score ranges from 0 (not at all impaired) to 35 (heavily impaired), with a cut-off for potential frailty at ≥6.
  Other Names: mG8
Diagnostic Test: 30 second chair stand test — Repetitions within 30 seconds
  Other Names: 30s-CST; chair stand test; 30 CST; CST; sit-to-stand test; 30 s chair stand test
Diagnostic Test: Handgrip Strength Test — Measured in kilograms
  Other Names: HGST; HST

SUMMARY:
Older patients with cancer constitute a heterogeneous group with varying comorbidity; therefore, geriatric assessment with initial screening is recommended. The Geriatric 8 (G8) has been established as a promising screening tool. Currently, there are no guidelines for oncogeriatric screening in older cancer patients in Denmark. We hypothesize that by screening persons age 70 years or more with newly diagnosed cancer, with the G8, we can assess the prognostic value and identify a subgroup of patients who will benefit from a CGA.

Aims:

* Determine whether Danish cancer patients, with a G8 score of ≤14, experience poorer quality of life (QoL), receive less recommended standard cancer treatment, experience more treatment-related toxicity, stop treatment earlier, and experience shorter survival than patients with a G8 score >14.
* Ascertain whether the standard G8 cut-off score of ≤14 is the most relevant cut-off score, with respect to treatment adherence, treatment-related toxicity, QoL, and survival, when focusing on the older Danish cancer patient population.
* Establish whether the performance and prognostic value of the G8 can be strengthened through the addition of a functional measure, the 30-second chair stand test (30-CST), and/ or the handgrip strength test (HGST).
* Evaluate the prognostic value of the modified Geriatric 8 (mG8)

Methods:

A prospective, descriptive study of all outpatients with newly diagnosed solid tumors at the Department of Oncology, Odense University Hospital, age 70 years or more. Patients will be screened with the G8, mG8, 30-CST, HGST, and QoL questionnaires at baseline with subsequent one-year follow-up, to determine the prognostic value of the G8 and the mG8. An initial two-month pilot study will help determine inclusion rates and highlight necessary practical adjustments to ensure optimal study participation. Baseline characteristics will be compared with descriptive statistics. Our primary endpoint; Global Health status/ QoL (EORTC QLQ-C30 & QLQ-ELD14), and secondary endpoints; treatment adherence, and treatment-related toxicity, will be assessed using logistical regression; while secondary endpoints; overall survival, cancer-specific survival, will be assessed using the Kaplan Meier analysis and Cox proportional hazard models. Post hoc diagnostic performance analysis will be conducted to determine the optimal G8 cut-off and whether functional measures (30-CST and HGST) can enhance screening accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥70 with solid tumors (not hematological malignancies nor non-melanoma skin cancer) referred to the outpatient clinic at Odense University Hospital for information and/or antineoplastic treatment
* Patients must be able to give informed consent
* Patients must be able to speak English or Danish

Exclusion Criteria:

* Patients who have received antineoplastic treatment for another cancer diagnosis within the past year
* Patients who have begun chemotherapy or immunotherapy for the referred cancer diagnosis, more than 48 hours prior to the time of consent
* Patients who have begun other antineoplastic treatment (not endocrine) for the referred cancer diagnosis, more than 7 days prior to the time of consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All outpatients, age 70 years or more with solid malignancies, referred to the Department of Oncology at Odense University Hospital for antineoplastic treatment or information
Sampling Method: Non-Probability Sample
Enrollment: 1401 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Global health status / Quality of Life | 12 months
  Global health status will be described using EORTC QLQ-C30

SECONDARY OUTCOMES:
Health-related Quality of Life (HRQoL) | 12 months
  HRQoL is measured by EORTC QLQ-C30
Health-related Quality of Life (HRQoL) | 12 months
  HRQoL is measured by EORTC QLQ-ELD14 (ELderly Cancer Patients Module)
Overall Survival | 12 months
  Overall Survival is measured from Geriatric 8 screening to time of death
Cancer-specific Survival | 12 months
  Cancer-specific Survival is measured from Geriatric 8 screening to time of death in patients with residual cancer
Adherence to initial oncologic treatment plan | 12 months
  Deviation from initial oncologic treatment plan with the registration of dose reductions, with the given dose measured as a percentage of the planned dose.
Adherence to initial oncologic treatment plan | 12 months
  Deviation from initial oncologic treatment plan with the registration of dose delays, measured in days.
Adherence to initial oncologic treatment plan | 12 months
  Deviation from initial oncologic treatment plan with the registration of discontinuation of treatment, measured as the number of given cycles divided by the number of planned cycles.
Performance analysis of the Geriatric 8 | 12 months
  Performance analysis will be conducted using patients allocated to Comprehensive Geriatric Assessment (CGA), where an abnormal CGA will be defined as >1 abnormal domain, in accordance with the Danish version of the Geriatric Core Dataset (G-Code).

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Ewertz, MD, DMSc, Study Director — University of Southern Denmark; Jesper Ryg, MD, PhD, Study Chair — Department of Geriatric Medicin, Odense University Hospital; Cecilia M Lund, MD, PhD, Study Chair — Department of Clinical Medicin, Herlev and Gentofte Hospital; Trine L Jørgensen, MD, PhD, Study Chair — Department of Oncology, Odense University Hospital; Per Pfieffer, MD, PhD, Study Chair — Department of Oncology, Odense University Hospital; Henrik J Ditzel, MD, DMSc, Study Chair — Department of Oncology, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ditzel HM, Giger AW, Lund CM, Ditzel HJ, Mohammadnejad A, Pfeiffer P, Ryg J, Jorgensen TL, Ewertz M. Predictive Value of Geriatric Oncology Screening and Geriatric Assessment in Older Patients with Solid Cancers: Protocol for a Danish prospective cohort study (PROGNOSIS-G8). J Geriatr Oncol. 2021 Nov;12(8):1270-1276. doi: 10.1016/j.jgo.2021.06.004. Epub 2021 Jun 25. PMID 34176752